CLINICAL TRIAL: NCT02476565
Title: Comparison of Endotracheal Intubation Over the Aintree Via the I-gel and Laryngeal Mask Airway Supreme
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Antonio Hernandez, Assoc Professor of Clinical Anesthesiology, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 131507
Record Dates: First submitted 2015-06-03; First posted 2015-06-19 (Estimated); Results first posted 2018-01-18 (Actual); Last update posted 2018-03-16 (Actual); Status verified 2018-02

CONDITIONS: Difficult Intubation
Keywords: Intubation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LMA-Supreme supraglottic device (Experimental): The LMA-Supreme is a single-use disposable supraglottic airway that utilizes an inflatable cuff
  Interventions: Device: LMA-Supreme supraglottic device
- I-gel supraglottic device (Active Comparator): The I-gel is an alternative supraglottic device made from thermoplastic elastomer which provides the seal over the airway versus an inflatable cuff.
  Interventions: Device: I-gel supraglottic device

INTERVENTIONS:
Device: LMA-Supreme supraglottic device — The fiberscope (with the Aintree loaded on top of it) will be advanced through the supraglottic device into the trachea. Next, the supraglottic device will be removed and the endotracheal tube will be advanced into the airway over the Aintree airway intubation catheter. Finally, the Aintree catheter is removed and the endotracheal tube will be left in the airway.
  Arms: LMA-Supreme supraglottic device
Device: I-gel supraglottic device — The fiberscope (with the Aintree loaded on top of it) will be advanced through the supraglottic device into the trachea. Next, the supraglottic device will be removed and the endotracheal tube will be advanced into the airway over the Aintree airway intubation catheter. Finally, the Aintree catheter is removed and the endotracheal tube will be left in the airway.
  Arms: I-gel supraglottic device

SUMMARY:
The investigators plan to conduct a randomized trial comparing the efficacy of intubating the tracheal using an Aintree intubation catheter through either the LMA-S or I-gel supraglottic devices

DETAILED DESCRIPTION:
With the proposal, the investigators are comparing two different types of supraglottic devices. One is the LMA Supreme (laryngeal mask airway) and the other is the I-gel. The study is designed to use the supraglottic airway device as an adjunct to tracheal intubation, not as the definitive airway. The investigators will be utilizing the Aintree intubation catheter over the fiberoptic bronchoscope in an effort to secure the airway. This technique has been well described in the literature and has been proven effective and safe.

ELIGIBILITY:
Inclusion Criteria:

* Subjects that will require routine endotracheal intubation for general anesthesia as part of their surgery.
* Age >18 years old.
* Can provide informed consent.

Exclusion Criteria:

* Subjects that require rapid sequence induction for endotracheal intubation; i.e., parturients, or any subject that is at high risk for aspirating gastric contents into the airway.
* Subjects that have an allergy to Propofol or eggs.
* Subjects that have an allergy to rocuronium.
* Subjects with a history of oropharyngeal or laryngeal surgery, or subjects undergoing oropharyngeal or laryngeal surgery.
* Subjects with congenital or anatomical airway anomalies.
* Subjects with anticipated reduced functional residual capacity as predicted by a body mass index ≥40.
* Currently enrolled in another research study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2014-09; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Hernandez, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (2):
- United States (2):
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - South Texas Veterans HealthCare System, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | I-gel Supraglottic Device | LMA-Supreme Supraglottic Device
Started | 20 | 19
Completed | 20 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LMA-Supreme Supraglottic Device | I-gel Supraglottic Device | Total
Number analyzed (Participants) | 19 | 20 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Data not available for 10 subjects
  years
    number analyzed (Participants) | 14 | 15 | 29
    (all) | 54 (15) | 58 (14) | 56 (14)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Data not available for 10 subjects
  Participants
    number analyzed (Participants) | 15 | 14 | 29
    Female | 1 | 2 | 3
    Male | 14 | 12 | 26
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19 | 20 | 39
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 28.3 (8.0) | 27.3 (8.3) | 27.7 (8.1)

OUTCOME MEASURES:

1. Primary Outcome: Time to Successful Tracheal Intubation
Description: This measure of time begins with the handling of the supraglottic device to confirming the appropriate placement of the device by noting the presences of end tidal carbon dioxide.
Time Frame: Up to 10 minutes
Population: unable to confirm accuracy of data in 1 participant in the I-gel group, that participant's data was not included in the analysis
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | I-gel Supraglottic Device | LMA-Supreme Supraglottic Device
Number analyzed (Participants) | 19 | 19
seconds | 197 (93) | 304 (173)

2. Secondary Outcome: Time to Placement of the Supra Glottic Device
Description: This measure of time begins with the handling of the supra glottic device to confirming the appropriate placement of the device by noting the presences of end tidal carbon dioxide
Time Frame: Up to 10 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | I-gel Supraglottic Device | LMA-Supreme Supraglottic Device
Number analyzed (Participants) | 19 | 19
seconds | 155 (182) | 301 (246)

3. Secondary Outcome: Percent of Subjects Who Required 0, 1, 2, and 3 Airway Manipulations for the Placement of the Supraglottic Device
Description: Percent of subjects who required 0, 1, 2, and 3 airway manipulations for the placement of the supraglottic device
Time Frame: Up to 10 minutes
Population: 4 participants in the LMA-Supreme arm were not included in analysis because the study was aborted at the request of the attending or the times to established safety cutoff for airway establishment (10 minutes) was exceeded.
Measure: Number; unit: percent of participants
Arm/Group | I-gel Supraglottic Device | LMA-Supreme Supraglottic Device
Number analyzed (Participants) | 20 | 15
percent of participants
  0 manipulations | 80 | 80
  1 manipulations | 10 | 13
  2 manipulations | 5 | 7
  3 manipulations | 5 | 0

4. Secondary Outcome: Time to Placement of the Aintree Airway Intubation Catheter
Description: This measure of time begins with the handling of the fiberscope to withdrawal of the fiberscope from the Aintree and setting the fiberscope down
Time Frame: Up to 10 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | I-gel Supraglottic Device | LMA-Supreme Supraglottic Device
Number analyzed (Participants) | 19 | 19
seconds | 155 (182) | 301 (246)

5. Secondary Outcome: Percent of Subjects Who Required 0, 1, 2, 3 and 6 Airway Manipulations for the Placement of the Aintree.
Description: Percent of subjects who required 0, 1, 2, 3 and 6 airway manipulations for the placement of the Aintree.
Time Frame: Up to 10 minutes
Population: 2 participants in I-gel arm were excluded from analysis because times to established safety cutoff for airway establishment(10 minutes) was exceeded. 3 participants in LMA-Supreme arm were excluded in analysis because study was aborted at request of attending or times to established safety cutoff for airway establishment (10 minutes) was exceeded.
Measure: Number; unit: percent of participants
Arm/Group | I-gel Supraglottic Device | LMA-Supreme Supraglottic Device
Number analyzed (Participants) | 18 | 16
percent of participants
  0 manipulations | 67 | 25
  1 manipulations | 33 | 25
  2 manipulations | 0 | 31
  3 manipulations | 0 | 12
  6 manipulations | 0 | 6

6. Secondary Outcome: Time to Placement of the Endotrotracheal Tube
Description: Time to the appropriate placement of the endotracheal tube.
Time Frame: Up to 10 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: second
Arm/Group | I-gel Supraglottic Device | LMA-Supreme Supraglottic Device
Number analyzed (Participants) | 19 | 19
second | 81 (71) | 96 (117)

7. Secondary Outcome: Percent of Subjects With 0, 1, 2 and 3 Airway Manipulations Required for Placement of Endotrachial Tube
Description: Percent of subjects with 0, 1, 2 and 3 airway manipulations required for placement of endotrachial tube
Time Frame: Up to 10 minutes
Population: 2 participants in I-gel arm were excluded from analysis because times to established safety cutoff for airway establishment(10 minutes) was exceeded. 5 participants in LMA-Supreme arm were excluded in analysis because study was aborted at request of attending or times to established safety cutoff for airway establishment (10 minutes) was exceeded.
Measure: Number; unit: percent of participants
Arm/Group | I-gel Supraglottic Device | LMA-Supreme Supraglottic Device
Number analyzed (Participants) | 18 | 14
percent of participants
  0 manipulations | 67 | 57
  1 manipulations | 17 | 43
  2 manipulations | 11 | 0
  3 manipulations | 6 | 0

8. Other Pre Specified Outcome: Visualization Score
Description: The visualization of each of the following structures provides one point, for a maximum score of 7.
  1. Right true vocal cord.
  2. Left true vocal cord.
  3. Right false vocal cord.
  4. Left false vocal cord.
  5. Right posterior cartilage
  6. Left posterior cartilage
  7. Epiglottis
Time Frame: Up to 10 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | I-gel Supraglottic Device | LMA-Supreme Supraglottic Device
Number analyzed (Participants) | 20 | 19
units on a scale | 6.0 (1.3) | 3.4 (2.9)

ADVERSE EVENTS:
Time Frame: from start of anesthesia to successful intubation, up to 10 minutes
Arm/Group | I-gel Supraglottic Device | LMA-Supreme Supraglottic Device
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/19
Other Adverse Events (participants affected / at risk) | 1/20 | 0/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | I-gel Supraglottic Device (N=20) | LMA-Supreme Supraglottic Device (N=19)
Coughing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Post Extubation Stridor (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes